CLINICAL TRIAL: NCT04193306
Title: ACAV: Efficacy and Safety Of Alirocumab to Prevent Early Cardiac Allograft Vasculopathy in Recent Heart Transplant Recipients
Brief Title: Efficacy and Safety Of Alirocumab to Prevent Early Cardiac Allograft Vasculopathy in Recent Heart Transplant Recipients
Acronym: ACAV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Vojtech Melenovsky, MD, PhD, Deputy director of the Research Department, senior consultant of the Heart Failure Division, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACAV2018
Record Dates: First submitted 2019-11-26; First posted 2019-12-10 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Allograft Vasculopathy
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded study with placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alirocumab (Experimental): alirocumab 150 mg s.c. every 2 weeks, for 48 weeks
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): placebo s.c. every 2 weeks, for 48 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alirocumab — Alirocumab 150 mg s.c. every 2 weeks
  Arms: Alirocumab
Other: Placebo — Placebo s.c. every 2 weeks
  Arms: Placebo

SUMMARY:
Cardiac allograft vasculopathy (CAV) represents the leading cause of late morbidity and mortality in heart transplant recipients as the second most frequent cause of all deaths at 3 years. In distinction from general coronary atherosclerosis, CAV affects diffusely the entire coronary vasculature with marked intimal proliferation and concentric vascular thickening and fibrosis. It was demonstrated that most of the intimal thickening due to CAV occurs during the first year after transplantation. Furthermore, the severity of the CAV appears to correlate with lipid abnormalities and elevated low-density lipoprotein cholesterol (LDL-C) is very common after transplantation with nadir of LDL levels occurring at 6 months.

Because of drug-drug interactions, heart transplant recipients cannot be treated with adequate doses of statins to achieve desirable reduction of LDL-C levels (reduction ˂ 60% of LDL-C). The use of alternative lipid-lowering drugs including bile acid sequestrates, fibrates, nicotinic acid or ezetimibe is not recommended in post-transplant scenario. Inhibition of proprotein convertase subtilisin/kexin type 9 (PCSK9) increase availability has emerged as a novel drug tool for LDL-C lowering, capable to lower LDL-C by more than 60% even in statin-treated patients with very good safety profile.

Although heart transplant recipients fulfill approved indication and standard clinical guidelines of a PCSK9 inhibitor, alirocumab, there are no available data on use of PCSK9 inhibitor in post-transplant situation.

The purpose of the ACAV study is to clarify efficacy and safety of alirocumab compared to placebo administered during the first year after transplantation in heart transplant recipients in addition to background atorvastatin therapy. Except lipid profile, optical coherence tomography (OCT) will be performed as the objective efficacy endpoint to examine thickness and lumen of coronary vessels. It is expected that inhibition of PCSK9 in heart transplant recipient will dramatically improve post-transplant lipoprotein levels and perhaps slow down development of CAV in the most critical period of the first year after transplantation.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, prospective, phase IV trial with parallel design. 126 of new cardiac transplant recipients are planned to be enrolled in two sites: 1) Transplant Centre at Institute for Clinical and Experimental Medicine, Prague, Czech Republic, and 2) St Anne's University Hospital (FNUSA) - Centre of Cardiovascular and Transplant Surgery (CKTCH) in Brno, Czech Republic. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. Screening period could last up to four weeks. Subjects will be randomized 1:1 to receive either alirocumab 150 mg every 2 weeks or placebo between month 1 and month 12 after transplantation (study treatment will start after the first surveillance cardiac catheterization approximately one month after heart transplantation and it will be completed after the second surveillance cardiac catheterization approximately 12 months after heart transplantation). Furthermore, all subjects will be on a background statin treatment with atorvastatin 10 mg daily. After Screening and Baseline visit, 5 visits are planned during the treatment period (4, 8, 20, 34 and 48 weeks after baseline) and follow-up visit is planned 60 weeks after baseline. Maximal expected duration of subject participation will be 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. New cardiac transplant recipient ≥ 18 years of age willing to participate in the study.
2. Ability to understand study procedures and to comply with them for the entire length of the study.
3. Written informed consent obtained from subject or subject's legal representative.
4. Heart transplantation surgery performed 3 - 8 weeks before the baseline visit.

Exclusion Criteria:

1. Known hypersensitivity/allergy reaction to study medication.
2. Complicated post-transplant outcome with poor neurological status, multiorgan failure or graft dysfunction.
3. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
4. Lipoprotein apheresis is planned of performed.
5. Level of LDL-C ≥ 8 mmol/L at screening.
6. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
7. Participation in any other interventional study.

Known hypersensitivity/allergy to contrast agent or severe renal insufficiency (eGFR ˂ 30 mL/min/1.75 m2) exclude patient from OCT imaging only, not from the whole study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
calculated LDL cholesterol concentration | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2,3,4,5 and 6 between alirocumab/placebo arms
HDL cholesterol concentration | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2,3,4,5 and 6 between alirocumab/placebo arms
total cholesterol | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2,3,4,5 and 6 between alirocumab/placebo arms
triglycerides | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2,3,4,5 and 6 between alirocumab/placebo arms
ApoB | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2,3,4,5 and 6 between alirocumab/placebo arms
Lp (a) | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2,3,4,5 and 6 between alirocumab/placebo arms
Apo A1 | the time period between 2 and 12 months after heart transplantation
  the difference in mean of values from visits 2, 3, 4 ,5 and 6 between alirocumab/placebo arms

SECONDARY OUTCOMES:
calculated LDL cholesterol concentration | between 1 and 12 months after heart transplantation
  Percent change from baseline (visit 1) to visit 6 between alirocumab/placebo arms
calculated LDL cholesterol concentration | between 1 and 12 months after heart transplantation
  Difference in values at every study visit between alirocumab/placebo arms
lipid parameters values | between 1 and 12 months after heart transplantation
  Difference in values at every study visit between alirocumab/placebo arms
calculated LDL cholesterol concentration | between 12 and 15 months after heart transplantation
  Difference in values at visit 6 compared to visit 7 between alirocumab/placebo arms
lipid parameters values | between 12 and 15 months after heart transplantation
  Difference in values at visit 6 compared to visit 7 between alirocumab/placebo arms
mean intimal thickness assessed by OCT | 1 and 12 months after heart transplantation
  Percent change from baseline (visit 1) to visit 6 between alirocumab/placebo arms
mean lumen volume assessed by OCT | 1 and 12 months after heart transplantation
  Percent change from baseline (visit 1) to visit 6 between alirocumab/placebo arms
incidence of adverse events | 1 and 15 months after heart transplantation
  Assessment of safety of alirocumab in comparison to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Z, Pazdernik M, Zhang H, Wahle A, Guo Z, Bedanova H, Kautzner J, Melenovsky V, Kovarnik T, Sonka M. Quantitative 3D Analysis of Coronary Wall Morphology in Heart Transplant Patients: OCT-Assessed Cardiac Allograft Vasculopathy Progression. Med Image Anal. 2018 Dec;50:95-105. doi: 10.1016/j.media.2018.09.003. Epub 2018 Sep 14. PMID 30253306
- [Background] Pazdernik M, Chen Z, Bedanova H, Kautzner J, Melenovsky V, Karmazin V, Malek I, Tomasek A, Ozabalova E, Krejci J, Franekova J, Wahle A, Zhang H, Kovarnik T, Sonka M. Early detection of cardiac allograft vasculopathy using highly automated 3-dimensional optical coherence tomography analysis. J Heart Lung Transplant. 2018 Aug;37(8):992-1000. doi: 10.1016/j.healun.2018.04.002. Epub 2018 Apr 6. PMID 29706574